CLINICAL TRIAL: NCT02625818
Title: The Genetic and Affective Prediction Study
Acronym: GAP
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/1751
Record Dates: First submitted 2015-12-04; First posted 2015-12-09 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Mental Disorders
Keywords: Emergency Services, Psychiatric; Prognosis; Biological markers; Anxiety; Panic; Psychomotor Agitation; Self-injurious Behavior
MeSH Terms: conditions — Mental Disorders; Anxiety Disorders; Psychomotor Agitation; Self-Injurious Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples (plasma and serum)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- acute psychiatric condition

SUMMARY:
A major proportion of patients admitted to psychiatric acute and emergency departments have symptoms, behaviors or function influenced by implicit or explicit suicidal intention (tendency towards self-harm, or suicide attempt). There is an increased risk of suicide in the acute phase during in-patient stay and after discharge. At present there is no satisfactory tool to predict post-discharge suicide risk.

Multidimensional rating is expected to have better predictive properties than one-dimensional rating for suicidal behavior during in -patient stay and two years after discharge. Multidimensional rating assesses anxiety, panic, agitation, suicidal thoughts and ideations, as well as therapist's reactions during interviews. In the present study the predictive properties of two rating scales for suicidal behavior during in-patient stay and two years after will be compared. One of these is a multidimensional scale: "Multidimensional Assessment of Suicide Risk" (MARIS).

ELIGIBILITY:
Inclusion Criteria:

* acute agitated condition
* informed consent

Exclusion Criteria:

* Drug abuse
* in-patient stay for a fixed time at regular intervals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the psychiatric acute department for central Norway, St Olavs University Hospital, Trondheim. The department has a catchment area of approximately 240000 inhabitants ≥ 18 years. The hospital has close to 2000 admittances each year
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
self-inflicted, potentially injurious behavior with intention to die defined as acts needing attendance by physician | 2 weeks
  during in-patient stay

SECONDARY OUTCOMES:
suicide | 2 years after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Randolf Terje Vågen, Study Director — St Olavs Hospital, Division of Mental Health Care; Nanna Sønnichsen Kayed, Study Director — Department of Mental Health, Faculty of Medicine and Health, NTNU
Locations (1):
- St Olavs Hospital, Østmarka psychiatric department, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No